CLINICAL TRIAL: NCT03487965
Title: A Randomized, Double Blinded, Placebo Controlled Clinical Study to Evaluate Skin Attributes Following Dietary Supplement Consumption
Brief Title: Evaluation of Skin Attributes Following Dietary Supplement Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Access Business Group (Industry)
Collaborators: Clinical Research Laboratories (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CRL119515
Record Dates: First submitted 2018-03-29; First posted 2018-04-04 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Skin Condition
Keywords: dicarbonyl compounds; skin elasticity; glycation
MeSH Terms: conditions — Skin Diseases | interventions — Polyphenols

STUDY DESIGN:
Intervention Model Description: individuals are assigned prospectively to two different interventions according to a protocol, to evaluate the effect of the interventions
Who Masked: Participant, Care Provider, Investigator
Masking Description: Interventions coded, blinded code kept in sealed envelope until study closed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Low dose Polyphenol (Experimental): 130 mg of Aronia Extract with 120 mg of licorice root combination blend provided to subjects once per day for 16 weeks.
  Interventions: Dietary Supplement: Low dose Polyphenol
- High dose Polyphenol (Experimental): 200 mg of Aronia extract provided to subjects once per day for 16 weeks
  Interventions: Dietary Supplement: High dose Polyphenol
- Placebo control (Placebo Comparator): Inert tablet provided to subjects once per day for 16 weeks
  Interventions: Dietary Supplement: Placebo Control

INTERVENTIONS:
Dietary Supplement: Low dose Polyphenol — botanical supplement with 25 mg polyphenol
  Arms: Low dose Polyphenol
Dietary Supplement: High dose Polyphenol — botanical supplement with 13 mg polyphenol
  Arms: High dose Polyphenol
Dietary Supplement: Placebo Control — inert tablet made to mimic the experimental tablets
  Arms: Placebo control

SUMMARY:
The study is to assess skin attributes of female subjects following 16 weeks of dietary supplement consumption.

DETAILED DESCRIPTION:
This is a 16 week, randomized, double blind, placebo controlled study. Approximately 105 Caucasian and Asian (Korean, Japanese, or Chinese) female subjects will be enrolled. The following clinical assessments will be performed: (1)VISIA-CR™ digital photography; (2)AGE Reader SU measurements on the left cheek and left inner forearm; (3) Visual Analog Grading (VAS); (4) Corneometer measurements; and (5) Cutometer measurements. Subjects will return to the clinic at approximately 4 weeks, 8 weeks and 16 weeks from the baseline visit for similar measurements. A self-perception questionnaire will be administered at the conclusion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a Caucasian or Asian (either Korean, Japanese, or Chinese) female between the ages of 30 and 65 years;
* Subject is overweight or moderately obese, with a BMI between 27 and 33;
* Subject is Caucasian and qualifies based on AGE Reader assessment that is at or greater than average for chronological age; OR is Asian and has an obtainable AGE Reader assessment on the left forearm. Screening AGE reader assessment will be done on the left inner forearm;
* Subject is willing to have fasting blood draws and urine collections at specified visits. At least nine hours fasting is required. Subject is allowed to drink water;
* Subject is willing to refrain from excessive sun exposure and/or the use of tanning beds;
* Subject is willing to use daily the provided facial SPF moisturizer and Purpose® cleansing bar;
* Subject is taking well established, stable doses of prescription and nonprescription medications not indicated to treat a thyroid condition or diabetes;
* Subject is in generally good health as determined by the medical history and blood panel results in the opinion of the Principal Investigator;
* Subject is dependable and able to follow directions as outlined in the protocol;
* Subject agrees to complete and sign a Photography Release Form, providing consent for the capture of facial digital images for use in relation to this clinical study;
* Subject has completed a HIPAA Authorization Form in conformance with 45 CFR Parts 160 and 164;
* Subject understands and is willing to sign an Informed Consent in conformance with 21 CFR Part 50: "Protection of Human Subjects."

Exclusion Criteria:

* Subject is pregnant, planning to become pregnant, or nursing;
* Subject is known to have, or at risk for, photosensitivity reactions (e.g. very sensitive to ultraviolet light);
* Subject has scars, tattoos, moles, age spots or rashes on the tested areas that the AGE Reader sensor and Cutometer® probe need to be placed;
* Subject takes prescription anticoagulants (this does not include a daily 81 mg dose of Aspirin);
* Subject has a history of any type of cancer and/or is currently undergoing treatment for any type of cancer;
* Subject has either a systolic blood pressure above 160 or a diastolic blood pressure above 100 at any time during the study;
* Subject has a thyroid condition;
* Subject is diabetic or taking any medication or herbal supplement to lower their blood glucose

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-04-28 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
Change of Skin Autofluoresence | Change from baseline to 16 weeks, change from 8 weeks to 16 weeks
  Change of accumulation of glycation as measured by validated autofluoresence measuring device (AGE Reader)

SECONDARY OUTCOMES:
Skin elasticity | Change from baseline to 16 weeks; change from 8 weeks to 16 weeks
  Relationship between elasticity and skin glycation; elasticity will be measured by cutometer

CONTACTS AND LOCATIONS:
Overall Officials: Anita L Cham, MD, Principal Investigator — Clinical Research Laboraties, LLC

IPD SHARING:
Plan to Share IPD: No